CLINICAL TRIAL: NCT00237211
Title: Study of High-dose Letrozole Therapy in Postmenopausal Patients With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFEM345F1201
Record Dates: First submitted 2005-10-09; First posted 2005-10-12 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Postmenopausal Women With Advanced Breast Cancer
Keywords: Aromatase inhibitor; letrozole; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

ARMS (1):
- Letrozole (Experimental)
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole
  Other Names: FEM345

SUMMARY:
To investigate the safety and efficacy of letrozole monotherapy at a dose of 2.5 mg/day in postmenopausal patients with breast cancer, and to determine the blood concentrations of letrozole and hormones.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically documented breast cancer.
* Patients with hormone receptor (ER and/or PgR) status of positive or unknown
* Patients who have been amenorrheic for the preceding 12 months or more.
* Patients who are 20 years or older and younger than 75 years.
* Patients with a history of postoperative adjuvant therapy or a history of endocrine therapy with tamoxifen for the treatment of progression or recurrence of the lesion. The endocrine therapy, however, should not exceed one regimen.
* Patients with progressing lesions.
* Patients with sufficient organ function to evaluate the safety
* Patients whose performance status (PS) is classified in 0～2.
* Patients who have no residual effects from previous treatments

Exclusion Criteria:

* Patients with other concurrent or previous malignant disease (excluding uterine carcinoma in-situ).
* Patients with hypercalcemia and uncontrollable cardiac disease (including a history of serious cardiac disease)
* Patients who have previously received aromatase inhibitor.
* Patients who have lymphangitis-type lung metastasis or symptomatic brain metastasis.

Other protocol-defined inclusion / exclusion criteria may apply.

Ages: 20 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2001-06; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Safety during treatment | Until disease progression or appearance of unacceptable toxicity whichever comes first
Response Rate during treatment | Until disease progression or appearance of unacceptable toxicity whichever comes first

SECONDARY OUTCOMES:
Pharmacokinetics measurement at baseline and at every 4 weeks until 28 weeks | Maximum 28 weeks after initiate treatment
Plasma estrogens level at baseline and at every 4 weeks until 28 weeks | Maximum 28 weeks after initiate treatment
Duration of response | From the first date of response confirmed and the last date of response confirmed
Time to progression | From the first date of response confirmed and the last date of response confirmed

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- Japan (12):
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, kooriyama, Fukushima
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Kitaadachi-gun, Saitama
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Fukushima
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Saitama